CLINICAL TRIAL: NCT04700410
Title: A New Method for Bowel Cleansing in Patients With a History of Poor Bowel Preparation - A Multicenter Feasibility Study With the Pure-Vu System
Brief Title: Bowel Cleansing Performance of the Pure-Vu System in Patients With a History of Poor Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: University Medical Center Mainz (Other); Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NL66613.091.18
Record Dates: First submitted 2020-12-17; First posted 2021-01-07 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer; Colonic Adenoma; Bowel Preparation
Keywords: Bowel preparation; colonoscopy; colorectal cancer; adenoma detection rate; endoscopy; therapeutic irrigation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: single arm international multicenter colonoscopy trial
Masking Description: Independent assessment of BBPS (photos).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pure-Vu (Experimental): All patients willing to participate will receive a limited bowel preparation (2-days of dietary restrictions + 2x 150ml picoprep) followed by intra-procedural bowel cleansing with the Pure-Vu System (single arm)
  Interventions: Device: Pure-Vu System

INTERVENTIONS:
Device: Pure-Vu System — All patients willing to participate will receive a limited bowel preparation (2-days of dietary restrictions + 2x 150ml picoprep) followed by intra-procedural bowel cleansing with the Pure-Vu System.

SUMMARY:
The diagnostic accuracy and safety of colonoscopy highly depends on the quality of the pre-procedural bowel preparation. A past history of poor bowel preparation is the most important risk factor of inadequate bowel cleansing at the next colonoscopy. This study aims to evaluate if an adequate level of bowel cleansing can be achieved with the Pure-Vu System in patients with previous poor bowel preparation, in a single arm international multicenter feasibility study.

DETAILED DESCRIPTION:
Rationale: It is widely acknowledged that the efficacy and safety of colonoscopy depends on the quality of the pre-procedural bowel preparation. Despite its importance, the proportion of colonoscopies with inadequate bowel preparation still ranges from 6.8-33% across studies. A past history of poor bowel preparation is the most important risk factor of inadequate bowel cleansing at the next colonoscopy. (1, 2) Evidence to recommend a specific bowel cleansing regimen in these patients is currently lacking. (3) Mostly, patients with previous bowel preparation are advised to drink more oral purgatives, which is very difficult and unpleasant for patients and therefore often fails.

The aim of this study is to evaluate if an intra-procedural bowel cleaning device, the Pure-VuTM System (Tirat Carmel, Israel) can be used to achieve an adequate level of bowel cleansing in patients with previous poor bowel preparation.

Objective: The aim of this study is to evaluate if an adequate level of bowel cleansing can be achieved with the Pure-Vu System in patients with previous poor bowel preparation (Boston Bowel Preparation Scale [BBPS]<6).

Study design: We will perform a single arm international multicenter colonoscopy trial. Adult patients with previous poor bowel preparation (BBPS<6) will be invited to participate in our study (n= 44). All patients willing to participate will receive a limited bowel preparation (2-days of dietary restrictions + 2x 150ml picoprep) followed by intra-procedural bowel cleansing with the Pure-Vu System. The BBPS will be assessed before and after segmental washing by the endoscopist who performs the procedure and later by an independent endoscopist (photos).

Study population: Adult patients with poor bowel preparation within the last 2 years. Exclusion criteria; previous colon resection, previous colorectal cancer, colitis, lower gastrointestinal bleeding with hemodynamic instability, ASA>3, insufficiently corrected anticoagulation disorders, inability to provide informed consent.

Primary endpoint: The primary endpoint of the study will be the BBPS-score before and after intra-procedural bowel cleaning with the Pure-Vu System.

Secondary endpoints include:

* Total number of colon lesions specified by histology
* Adenoma detection rate
* Cecal intubation rates
* Procedure times (total procedure time, cecal intubation time, withdrawal time, time for all other interventions)
* Total amount of water used for washing and total amount of fluids+residual stool removed.
* Patient reported outcomes (level of discomfort during bowel preparation and during colonoscopy on a visual analog scale)
* System usability
* Endoscopists' learning curve
* Safety outcomes

Nature and extent of the burden and risk associated with participation, benefit and group relatedness: Colonoscopy is a commonly performed procedure and the overall serious adverse event (SAE) rate is low, around 2.8 per 1000 colonoscopies. The risk of adverse events (AE) with the Pure-Vu are believed to be equivalent to conventional colonoscopy, including bleeding and perforation risks (13). Participation in this study could potentially benefit colonoscopy patients because the Pure-Vu is expected to improve the quality of colonoscopy. Inadequate bowel cleansing may be prevented by the Pure-Vu System. Inadequate bowel cleansing is associated with lower adenoma detection rates (ADR), lower completion rates, longer procedure times, more complications and a higher need for repeat procedures.(4, 5) In addition, Pure-Vu reduces the reliance on patients pre-procedural bowel preparation which is often considered the most deterrent part of colonoscopy by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18 and 80 years, referred and scheduled for either screening, diagnostic, or surveillance colonoscopy.
* Poor bowel preparation within the last 2 years, defined as a BBPS <6 or need for repeat colonoscopy or shortening of surveillance interval due to poor bowel preparation

Exclusion Criteria:

* Prior colon resection
* Previous colorectal cancer
* Colitis
* Lower gastrointestinal bleeding with hemodynamic instability
* Bowel obstruction
* Pregnancy or lactating
* ASA > 3
* Insufficiently corrected anticoagulation disorders
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation scale (BBPS)-score before cleaning with the Pure-Vu system. | 1 day (day of intervention)
  Boston Bowel Preparation scale (BBPS): The adequacy of bowel preparation should be assessed after all appropriate efforts to clear residual debris is completed. All three bowel regions of the colon will be scored (i.e., the right colon, transverse colon, and left colon) from 0-3 points by the endoscopist. The segment scores are summed for a total BBPS ranging from 0 to 9. The points will be assigned as follows:
  0) Unprepared colon segment with mucosa not seen because of solid stool that could not be cleared.
  1. Portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen because of staining, residual stool, and/or opaque liquid.
  2. Minor amount of residual staining, small fragments of stool, and/or opaque liquid but mucosa of colon segment seen well.
  3. Entire mucosa of colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid. Each segment of the colon received a segmental score from 0- 3.
Boston Bowel Preparation scale (BBPS)-score after cleaning with the Pure-Vu system. | 1 day (day of intervention)
  Boston Bowel Preparation scale (BBPS): The adequacy of bowel preparation should be assessed after all appropriate efforts to clear residual debris is completed. All three bowel regions of the colon will be scored (i.e., the right colon, transverse colon, and left colon) from 0-3 points by the endoscopist. The segment scores are summed for a total BBPS ranging from 0 to 9. The points will be assigned as follows:
  0) Unprepared colon segment with mucosa not seen because of solid stool that could not be cleared.
  1. Portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen because of staining, residual stool, and/or opaque liquid.
  2. Minor amount of residual staining, small fragments of stool, and/or opaque liquid but mucosa of colon segment seen well.
  3. Entire mucosa of colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid. Each segment of the colon received a segmental score from 0- 3.

SECONDARY OUTCOMES:
Total number of colon lesions specified by histology | 1 day (day of intervention)
Adenoma detection rate | 1 day (day of intervention)
Cecal intubation rates | 1 day (day of intervention)
Procedure times (total procedure time, cecal intubation time, withdrawal time, time for all other interventions) | 1 day (day of intervention)
Total amount of water used for washing and total amount of fluids+residual stool removed. | 1 day (day of intervention)
Patient reported outcomes (level of discomfort during bowel preparation and during colonoscopy on a visual analog scale) | 1 month
  A visual analogue scale from 0 to 10, in which higher numbers indicate a higher level of discomfort.
System usability | through study completion, an average of 1 year
  general ease of use, ease of rectum insertion, ease of angulation, ease of advancement, device stiffness, ease of polyp resection holding forces, ease of retroflexion,
  * Unacceptable
  * Difficult
  * Acceptable
  * Good (as good as conventional colonoscopy)
  * Excellent
Endoscopists' learning curve | through study completion, an average of 1 year
Number of adverse events after study intervention | 48 hours and 1month after intervention
  Safety outcomes (adverse events): Severe adverse events will be subcategorized cardiac (cardiac ischemia, heart failure, arrhythmia, other) pulmonary (exacerbation of Chronic Obstructive Pulmonary Disease, infectious, other), neurological (stroke, cerebrovascular accident, bleeding, other), and other (surgical interventions etc.).

CONTACTS AND LOCATIONS:
Locations (2):
- University Medical Center Mainz, Mainz, Germany
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Access Criteria: Data will be shared upon reasonable request